CLINICAL TRIAL: NCT01240174
Title: Demonstration of Near Zero Antibiotic Prescribing for Acute Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey A. Linder, Associate Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P001247
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Bronchitis; Cough
Keywords: Antibiotic; Antimicrobial; Prescribing; Cough; Acute Bronchitis
MeSH Terms: conditions — Bronchitis; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Arm (Other): Single arm in the study of doctors receiving feedback about their antibiotic prescribing rate for acute bronchitis.
  Interventions: Behavioral: Demonstration of near zero antibiotic prescribing for patients with acute bronchitis

INTERVENTIONS:
Behavioral: Demonstration of near zero antibiotic prescribing for patients with acute bronchitis — A controlled, continuously-monitored, implementation of an EHR-integrated diagnosis and treatment algorithm for acute bronchitis in a large, diverse primary care practice.

SUMMARY:
Studies show, guidelines state, and performance measures assert that antibiotic prescribing for uncomplicated acute bronchitis is inappropriate. However, clinicians prescribe antimicrobials in over 60% of the 22.5 million acute bronchitis visits in the United States each year. Previous successful interventions have only reduced the antimicrobial prescribing rate to 40% or 50%. It is unknown if the antimicrobial prescribing rate for acute bronchitis can be brought to near zero percent in actual practice while maintaining patient safety and satisfaction. The goal of this study is to develop an Electronic Health Record (EHR)-integrated algorithm for the diagnosis and treatment of adults with acute bronchitis with a goal of reducing the antibiotic prescribing rate to near zero percent.

DETAILED DESCRIPTION:
We will use a multi-modal implementation - including computerized decision support, reporting tools, and clinician feedback - and quality improvement techniques to ensure adherence to the algorithm and reduce the antimicrobial prescribing rate to near zero percent. The duration of the intervention will be 4 years.

ELIGIBILITY:
Inclusion Criteria:

* first visit in 30 days, age 18-64, has a cough of less than 3 weeks duration

Exclusion Criteria:

* infiltrate on chest x-ray, has chronic lung disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing rate | 30 days
  The antibiotic prescribing rate for patients with acute bronchitis

SECONDARY OUTCOMES:
Patient symptoms | 21 days
Patient satisfaction | 21 days
Patient safety | 30 days
Healthcare costs | 30 days
The capture and description of the components that had the greatest effect on the antimicrobial prescribing rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Linder, MD, MPH, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital Jen Center for Primary Care, Boston, Massachusetts, United States